CLINICAL TRIAL: NCT06847321
Title: A Randomized, Double-Blind, Placebo-Controlled Study of LHP588 in Subjects With P. Gingivalis-Positive Alzheimer's Disease
Brief Title: Study of LHP588 in Subjects With P. Gingivalis-Positive Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lighthouse Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LHP588-201
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Alzheimer Disease Due to P. Gingivalis
Keywords: placebo-controlled; p. gingivalis; Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Drug
- LHP588 25 mg (Experimental)
  Interventions: Drug: LHP588
- LHP588 50 mg (Experimental)
  Interventions: Drug: LHP588

INTERVENTIONS:
Drug: LHP588 — 25 mg
  Other Names: Low dose
  Arms: LHP588 25 mg
Drug: LHP588 — 50 mg
  Other Names: High dose
  Arms: LHP588 50 mg
Drug: Placebo Drug — Placebo
  Arms: Placebo

SUMMARY:
This study is to test LHP588 in persons who have mild to moderate Alzheimer's disease (AD) who have shown progressive mental decline in the last year and who have P. gingivalis infection. P. gingivalis infection has been linked to the development of dementia. LHP588 is designed to target the P. gingivalis bacterium, to potentially help to halt or slow down the progression of AD and its symptoms. A saliva test will be done to determine P. gingivalis infection. Tests for AD include standard questionnaires such as MMSE and a blood test for pTau 217. Treatment will be blinded, meaning the participant and the doctor will not know if the participant is receiving LHP588 or placebo. The total time for participation in the study may be up to 64 weeks. This includes a screening period (to ensure the participant is suitable for the study and the study is suitable for the participant) of up to 12 weeks, a treatment period of up to 48 weeks, and a safety follow-up period of 4 weeks after the last dose of the study drug to check the participant's overall health. Treatment is a once-a-day capsule. Caregiver participation is required. The study requires the participant to visit the study center (with the caregiver) at least 20 times within 64 weeks (this does not include any unplanned visits that may be recommended by the study doctor). In addition, the study doctor or clinic staff will contact the participant via phone at least 1 time.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study that will assess the efficacy and safety of LHP588 in participants with evidence of P. gingivalis [Pg] infection and Alzheimer's Disease (AD) according to the National Institute on Aging-Alzheimer's Association (NIA-AA) research criteria. Enrolled participants must also have evidence of P. gingivalis infection as determined by polymerase chain reaction (PCR) of saliva oral rinse and clinical evidence of progressive cognitive decline in the last year. The participant should not have other conditions or brain imaging abnormalities that can explain the symptoms of dementia based on prior imaging and the screening magnetic resonance imaging (MRI). Due to the nature of AD, participants must identify a primary caregiver prior to enrollment in the study who will assist the participant with study participation and attend clinic visits.

The study will consist of the following periods: 1) screening period of up to 12 weeks, 2) double-blind treatment period of 48 weeks (including a 2 week up-titration for the high dose arm), and 3) safety follow-up period of 4 weeks.

The screening period will include at least two office visits during which eligibility will be verified. The first screening visit assessments will be limited to only include the Mini-Mental State Examination (MMSE) and a saliva sample collection to assess P. gingivalis positivity for participants with the MMSE score of 12 to 24, inclusive. The second screening visit will only be scheduled for participants with positive results of Pg infection test and the rest of the screening procedures will be performed. Screening MRI will be performed as the last eligibility verification assessment.

Participants who meet all eligibility criteria will be randomized in a 1:1:1 fashion to receive LHP588 25 mg, LHP588 50 mg, or placebo, orally, once daily (QD) in a fasted state (at least one hour before or two hours after a meal) for 48 weeks. Dosing should be done at approximately the same time each day. Blood samples for pharmacokinetics levels and biomarkers will be collected during selected visits.

Evaluations will be conducted according to the schedule of assessments and will include: Medical history, physical examination, height, weight, saliva rinse for verification of P. gingivalis infection, Modified Hachinski, urine drug screen, magnetic resonance imaging (MRI) or computed tomography (CT) of the brain, Mini-Mental State Examination (MMSE), Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog 11), Alzheimer's Disease Cooperative Study Group-Activities of Daily Living (ADCS-ADL), Clinical Dementia Rating-Sum of Boxes (CDR-SB), blood for pharmacokinetic analysis, safely laboratory measures, electrocardiogram, Columbia-Suicide Severity Rating Scale (C-SSRS), and other tests or assessments.

After completion of study treatment, participants will continue to be monitored for 4 weeks and will have a phone call to assess safety at Week 50 and will return for the Safety Follow-up Visit (Week 52).

ELIGIBILITY:
Inclusion Criteria:

* AD according to the National Institute on Aging-Alzheimer's Association criteria.
* MMSE score between 12 and 24.
* Saliva rinse sample positive for P. gingivalis.
* Plasma pTau217 above cutoff.
* Subject and caregiver have provided full written informed consent.
* Background symptomatic therapy with acetylcholinesterase inhibitors, and/or memantine, are allowed if the dose has been stable for 90 days and no changes are planned during the study.
* Modified Hachinski score ≤4 at screening.

Exclusion Criteria:

* History of cancer requiring systemic therapy in last 5 years.
* Evidence of a clinically significant, unstable cardiovascular, pulmonary, renal, hepatic, gastrointestinal, neurologic, or metabolic disease within 6 months prior to screening.
* Unstable angina, uncompensated and/or symptomatic congestive heart failure (Grade 2 or higher on the New York Heart Association scale) or myocardial infarction within 6 months.
* Acute or poorly controlled blood pressure >180 mmHg systolic or >100 mmHg diastolic at screening visit.
* History or current evidence of major neurological or psychiatric illness such as schizophrenia, bipolar disorder, Parkinson's Disease, other.
* Currently being treated with anti-amyloid beta antibodies or other disease-modifying treatments for dementia.
* Other criteria in the Investigator's judgement that may interfere with the ability to participate in the study.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ADAS-Cog11 to the end of treatment period (at Week 40 - 48) | 40 - 48 weeks

SECONDARY OUTCOMES:
Change from baseline in CDR-SB to the end of treatment (at Week 40-48) | 40 - 48 weeks
  Clinical Dementia Rating-Sum of Boxes
Change from baseline in ADCS-ADL to the end of treatment (at Week 40-48) | 40 - 48 weeks
  Alzheimer's Disease Cooperative Study Group-Activities of Daily Living

CONTACTS AND LOCATIONS:
Locations (1):
- Northwest Clinical Research Center, Bellevue, Washington, United States

IPD SHARING:
Plan to Share IPD: No